CLINICAL TRIAL: NCT03850223
Title: Clinical Audit On Management Of Congenital Heart Disease In Assiut Children University Hospital
Brief Title: Clinical Audit On Management Of Congenital Heart Disease In ACUH
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Fadwa Magdy Mohamed Abdou, Principle investigator, Assiut University
Other Study IDs: MOCHD
Record Dates: First submitted 2019-02-20; First posted 2019-02-21 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Congenital Heart Disease (CHD) is the most common birth defect in the United States, affecting approximately 0.8% of live births. Improved treatment strategies and interventions have increased survival such that 85% to 90% of affected children are expected to live well into adulthood, thereby causing a demographic shift in which adults now outnumber children with CHD, and more people with complex CHD are living longer.

DETAILED DESCRIPTION:
CHD may be defined as an anatomic malformation of the heart or great vessels which occurs during intrauterine development, irrespective of the age at presentation. The cause of most congenital heart defects is still unknown. Many cases of congenital heart disease are multifactorial and result from a combination of genetic predisposition and an environmental stimulus. A small percentage of congenital heart lesions are related to known chromosomal abnormalities, in particular, trisomy 21, 13, and 18 and Turner syndrome. Of all cases of congenital heart disease, 2-4% are associated with known environmental or adverse maternal conditions and teratogenic influences, including maternal diabetes mellitus, phenylketonuria, systemic lupus erythematosus or congenital rubella syndrome; and maternal ingestion of drugs (lithium, ethanol, warfarin, antimetabolites, vitamin A derivatives, anticonvulsant agents).

ELIGIBILITY:
Inclusion Criteria:

* children with CHD more than one month

Exclusion Criteria:

* children with CHD less than one month

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children with congenital heart disease more than one month and less than 18 years
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2021-10-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Clinical audit study to assess management of congenital heart disease in AUCH | One year
  To assess how much the adopted protocol of management of congenital heart disease is implemented in Assiut university children hospital